CLINICAL TRIAL: NCT07283315
Title: Exploratory Clinical Study on the Safety and Efficacy of Second-generation CD19/BCMA Chimeric Antigen Receptor NK Cell Injection in Treating Paediatric B Cell-related Autoimmune Diseases
Brief Title: Exploratory Clinical Study of Second-generation CD19/BCMA Chimeric Antigen Receptor NK Cell Injection in Treating Paediatric B Cell-related Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Rui Therapeutics (Unknown)
Responsible Party: Principal Investigator, Mao Jianhua, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SC-0007-P-01
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Paediatric B Cell-related Autoimmune Diseases; Autoimmune Diseases; CAR
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/BCMA CAR NK cells (Experimental)
  Interventions: Biological: anti-CD19/BCMA CAR NK cells (KN5601-K)

INTERVENTIONS:
Biological: anti-CD19/BCMA CAR NK cells (KN5601-K) — The study adopted a dose-escalation and expansion study design. All subjects will receive fludarabine/ cyclophosphamide lymphodepletion followed by anti-CD19/BCMA CAR NK cells infusion.

SUMMARY:
Evaluating the efficacy and safety of anti-CD19/BCMA CAR-NK Cells in Paediatric B cell-related autoimmune diseases

ELIGIBILITY:
Inclusion Criteria:

* Common Inclusion Criteria:

  1. Informed consent: The participant (and guardian if the participant is a minor) must provide written informed consent, indicating understanding of the study purpose and procedures and willingness to participate.
  2. Cardiac Function: Echocardiography shows no significant structural abnormalities and left ventricular ejection fraction (LVEF) ≥ 55%.
  3. Hepatic Function: ALT ≤ 3 × ULN (except when elevation is attributable to inflammatory myopathy); AST ≤ 3 × ULN (except when elevation is attributable to inflammatory myopathy); Total bilirubin ≤ 2.0 × ULN (≤ 3.0 × ULN allowed for Gilbert syndrome).
  4. Renal Function: eGFR ≥ 30 mL/min/1.73 m².(Participants with eGFR < 30 mL/min/1.73 m² and/or those receiving renal replacement therapy may be considered eligible if, in the investigator's judgment, the potential benefit outweighs the risk and the participant or guardian provides fully informed consent.)
  5. Pulmonary Function: No severe pulmonary disease, and SpO₂ ≥ 92%.
  6. Women of childbearing potential must use medically acceptable contraception or practice abstinence during the study treatment period and for at least 12 months after the end of study treatment.

Disease-Specific Inclusion Criteria

SLE:

1. Age ≥ 5 years.
2. Meets the 2012 SLICC or 2019 EULAR/ACR classification criteria for SLE.
3. Must meet at least one of the following adequate treatment conditions:

   1. Treated with glucocorticoids (≥1 mg/kg/day prednisone or equivalent) plus one or more immunomodulatory agents (including cyclophosphamide, MMF, azathioprine, methotrexate, cyclosporine, tacrolimus, sirolimus, leflunomide, thalidomide, belimumab, or rituximab) for at least 3 months.
   2. Patients unable to tolerate conventional therapy may be eligible if, in the investigator's judgment, the potential benefit outweighs the risk and the participant (or guardian if minor) provides fully informed consent.
   3. Patients who cannot taper glucocorticoids to ≤5 mg/day after 6 months of conventional therapy.
4. SLE disease activity: SLEDAI-2K score ≥ 6.
5. No occurrence of macrophage activation syndrome within 1 month prior to screening.

MDR-SRNS

1. Age ≥3 years old, male or female.
2. Diagnosed with SRNS according to the 2021 Kidney Disease: Improving Global Outcomes #KDIGO# Guidelines;
3. Must meet at least one of the following adequate treatment conditions:

   1. have not achieved a complete response after 12 months of treatment with two standard doses of hormone replacement drugs with different mechanisms of action or relapse of disease activity after remission(at least one of the two drugs is a calcineurin inhibitor such as cyclosporine or tacrolimus, Other replacement drugs include Mycophenolate Mofetil, cyclophosphamide, Taitacept or rituximab).
   2. if no remission has been achieved after 3 to 6 months of adequate treatment with one calcineurin- inhibitor. The researcher judges that the benefits outweigh the risks and the patient or guardian has fully informed consent, the patient can be considered for inclusion.
   3. Patients with other diseases, such as systemic lupus erythematosus, requiring long-term systemic treatment with glucocorticoids or immunosuppressants, may be considered for inclusion after the investigator determines that the benefits outweigh the risks, and the patient or guardian has fully informed consent.
   4. Patients unable to tolerate conventional therapy may be eligible if, in the investigator's judgment, the potential benefit outweighs the risk and the participant (or guardian if minor) provides fully informed consent.
4. Renal biopsy was performed and the pathological type was determined to be minimal lesion nephropathy(MCD) or focal segmental glomerulosclerosis (FSGS);

IgA nephropathy

1. Age: ≥ 5 years old,male or female;
2. IgA nephropathy pathologically confirmed by renal biopsy;
3. Angiotensin-Converting Enzyme Inhibitors (ACE) or angiotensin receptor blocker (ARB) treated for at least 3 months and meet at least one of the following requirements:

   1. Combination or sequential treatment with steroids and at least one immunosuppressant or biologic for ≥ 3 months; and 24-hour urine protein quantification ≥500mg or UPCR≥0.5mg/mg;
   2. >50% decline in eGFR within 3 months;
   3. Patients who are unable to tolerate conventional treatment and for whom the investigator determines the benefits outweigh the risks and who have obtained fully informed consent from the patient or guardian may be considered for inclusion;
4. Exclude subjects with other secondary causes; exclude patients with uncontrolled blood pressure.

Refractory/Relapsed/Progressive Systemic Sclerosis:

1. Age: ≥ 5 years old, male or female;
2. Scleroderma fulfilling the 2013 ACR classification criteria
3. Positive scleroderma-related antibodies.
4. Modified Rodnan Skin Score (mRSS) ≥ 15 (total score 51).
5. Must meet at least one of the following adequate treatment conditions:

   1. Treated with glucocorticoids (≥0.5 mg/kg/day) plus at least one immunomodulatory agent (including antimalarials, cyclophosphamide, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, or biologics such as rituximab, belimumab, thalidomide) for more than 3 months without significant improvement.
   2. Meets criteria for rapidly progressive disease (see Appendix 1) and is unresponsive to standard therapy; participant may be enrolled if the investigator determines that potential benefit outweighs risk and informed consent is obtained.
   3. Patients unable to tolerate conventional therapy may be eligible if the investigator determines that potential benefit outweighs risk and informed consent is obtained.
6. Presence of severe pulmonary arterial hypertension (PAH), defined as a mean pulmonary arterial pressure >45 mmHg, or other severe involvement of major organs will be exclude.

Refractory/Relapsed ANCA-Associated Vasculitis:

1. Age: ≥ 5 years old, male or female;
2. Meets the diagnostic criteria for ANCA-associated vasculitis according to the 2007 European Medicines Agency (EMA) algorithm or the 2022 ACR/EULAR classification criteria, including microscopic polyangiitis (MPA) and granulomatosis with polyangiitis (GPA).
3. Has received glucocorticoids (≥1 mg/kg/day) in combination with at least one immunosuppressant or biologic agent (including cyclophosphamide, rituximab, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, belimumab, telitacicept, etc.) for at least 3 months without achieving sustained remission, or has experienced relapse after remission;or meets the criteria for severe vasculitis (Appendix 1), with inadequate response to standard-of-care therapy, and may be considered for enrollment if the investigator determines that the potential benefits outweigh the risks and the patient or legal guardian provides fully informed consent.
4. Evidence of active vasculitis meeting the following criteria: For participants <18 years of age: Pediatric Vasculitis Activity Score (PVAS) ≥10 (total score 63); For participants ≥18 years of age: Birmingham Vasculitis Activity Score (BVAS) ≥10 (total score 63); indicating active vasculitis.
5. Exclusion Criterion: Presence of alveolar hemorrhage requiring ventilatory support for more than one week.

Exclusion Criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, tocilizumab), or subjects with a history of severe allergic reactions.
2. Uncontrollable infection, or active infection that requires systemic treatment at screening.
3. Subjects with grade III or IV heart failure (NYHA classification).
4. Have a history of congenital heart disease or acute myocardial infarction within 6 months prior to screening; Or severe arrhythmias (including multisource frequent supraventricular tachycardia, ventricular tachycardia, etc.); Or combined with moderate to massive pericardial effusion, serious myocarditis, etc; Or patients with unstable vital signs who need hypertensive drugs.
5. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive; Or cytomegalovirus (CMV) DNA test positive.
6. History of severe herpes infection prior to screening, such as herpetic encephalitis, ocular herpes, or disseminated herpes; Signs of herpes or varicella-zoster virus infection (especially chickenpox, shingles) within 12 weeks prior to screening.
7. Patients with active central nervous system disease.
8. Patients with malignant diseases such as tumors before screening.
9. Secondary or congenital immunodeficiency.
10. History of any cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal disease or other major medical condition that would prevent the administration of KN5601-K, except for lupus.
11. Received solid organ transplantation or hematopoietic stem cell transplantation within 3 months prior to screening; Acute graft-versus host disease (GVHD) of grade 2 or above was present within 2 weeks prior to screening.
12. Received live vaccine within 4 weeks before screening.
13. Tested positive in Blood pregnancy test.
14. Patients who had participated in other clinical trials and received any intervention within 3 months before enrollment.
15. Any abnormal laboratory test results judged by the investigator to be clinically significant and prevent the subject from participating in the study. Laboratory test values that are out of range and not of clinical significance will not be considered as exclusion criteria.
16. Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicity (DLT) and treatment-emergent adverse events (TEAEs) | 1 month
  The safety of CAR-NK cell therapy in patients with B cell mediated autoimmune disease
response rate | 3 month
  The Efficacy of CAR-NK cell therapy in patients with SLE, MDR-SRNS, IgA nephropathy, or ANCA-AAV
CRISS score | 3 month
  The Efficacy of CAR-NK cell therapy in patients with Systemic Sclerosis

SECONDARY OUTCOMES:
Complete response or partial response rate | 6 month
  The Efficacy of CAR-NK cell therapy in patients with SLE, MDR-SRNS, IgA nephropathy, or ANCA-AAV, SSC

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No